CLINICAL TRIAL: NCT02532738
Title: A Stage II Clinical Trial Comparing the Efficiacy of Routine Treatment Combined With or Without MSC Therapy in Refractory Crohn's Disease
Brief Title: The Efficiency of MSC in Refractory Crohn's Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSCINRCD
Record Dates: First submitted 2015-08-23; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Crohn's Disease
Keywords: efficacy of MSC; refractory
MeSH Terms: conditions — Crohn Disease | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MSC-1 (Experimental): Patients in this arms receive routine treatment with 3×10E6/kg of MSC
  Interventions: Drug: Routine Treatment of CD; Biological: MSC treatment 01
- MSC-2 (Experimental): Patients in this arms receive routine treatment with 6×10E6/kg of MSC
  Interventions: Drug: Routine Treatment of CD; Biological: MSC treatment 02
- Ctrl (Placebo Comparator): Patients in this arms receive routine treatment with NS injection
  Interventions: Drug: Routine Treatment of CD; Other: NS

INTERVENTIONS:
Drug: Routine Treatment of CD — The Drug including 6MP, AZA, infliximab and thalidomide
Biological: MSC treatment 01 — Injection of 3×10E6/kg of MSC
  Arms: MSC-1
Biological: MSC treatment 02 — Injection of 6×10E6/kg of MSC
  Arms: MSC-2
Other: NS — Injection of NS
  Other Names: normal saline
  Arms: Ctrl

SUMMARY:
The investigators' preliminary study indicates that MSC is effective therapy in treating IBD. But the standard treatment is still lacking and the effect is not stable in IBD patients. This study is to explore the efficacy and standard strategy when using MSC in refractory IBD.

ELIGIBILITY:
Inclusion Criteria:

* Failure or intolerance to GC, immune inhibitors and biological agents treatment
* CDAI between 250-450
* Weight between 40-150 kg
* Normal renal function
* endoscopic or imaging diagnosis of CD in the small intestine, colon ileocolon
* Signed informed consent

Exclusion Criteria:

* HIV or active hepatitis patients;
* Allergic to CT contrast agents, cattle or pig products;
* Stricture or perforation type CD;
* Recieved permanent colostomy;
* Used biological preparation in 3 months
* Used prednisone > 20 mg/day within 1 month ;
* Patients with short bowel syndrome;
* Need total parenteral nutrition;
* Liver meritorious service is abnormal;
* Suffering from malignant tumor during the last 5 years;
* Combined bacterial or viral enteritis;
* Suffering from intestinal typicality thickening of the living
* Patients with tuberculosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Response of CD patients 12 weeks after receiving treatment (Reduction of CDAI score at less 100) | 12 weeks after receiving treatment
  Reduction of CDAI score at less 100

SECONDARY OUTCOMES:
Clinical Response of CD patients 6 weeks after receiving treatment (CDAI score less than 150) | 6 weeks after receiving treatment
  CDAI score less than 150